CLINICAL TRIAL: NCT05052658
Title: Time for Neuraxial Block Placement With Use of Ultrasound in Patients With High BMI
Brief Title: Ultrasound High BMI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Regina Fragneto, Professor, Dept of Anesthesiology, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69690
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Obesity Complicating Childbirth
Keywords: High BMI, pregnancy, ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palpation Group (Active Comparator)
  Interventions: Procedure: Neuraxial block placement
- Ultrasound Group (Experimental)
  Interventions: Procedure: Neuraxial block placement

INTERVENTIONS:
Procedure: Neuraxial block placement — The time and ease of administering neuraxial blocks in high BMI patients,for the management of labor and delivery pain, will be assessed.

SUMMARY:
This is a prospective experimental pilot study of full-term non-emergent obese parturients whose labor is being managed with epidural anesthesia to determine if neuraxial block placement with pre-procedure handheld ultrasound affects time to placement or number of needle passes. Approximately 25 patients, presenting for delivery at the University of Kentucky HealthCare Obstetrics Department, will be randomized to either the ultrasound or palpation group, between study approval and 31 July 2022.

DETAILED DESCRIPTION:
Placement of neuraxial blocks is commonly achieved by palpating surface landmarks. This somewhat "blind" technique to identify the spinal space becomes more difficult and less reliable in obese patients. Ultrasound devices have become common and successful with blocks and venous access, both involving mostly soft tissues. Application of conventional ultrasound for neuraxial blocks has been limited by its bulkiness, limited imaging for bony structures and a long learning curve. A newly developed pocket-size ultrasound addresses these limitations by providing real-time pattern recognition for spinal bony structures and 3D overlay for recognition of midline spinous process and intervertebral space using an automated artificial intelligent algorithm. The hypothesis is that ultrasound guidance will reduce time to epidural placement and reduce number of passes in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject requesting and consenting for a labor epidural, aged 18-50 and BMI between 35-59.9 at admission for labor.
* Subject with American Society of Anesthesiologists score equal to or less than III.
* Subject with singleton gestation equal to or greater than 37 weeks.
* Subjects with planned labor epidural in sitting position.

Exclusion Criteria:

* Patients with urgent or emergent diagnoses involving the health of the patient or child, such as abnormal fetal heart tracing.
* Patients with major back abnormalities (back surgery, significant scoliosis).
* Patients with contra-indication to neuraxial block (bleeding risk, local anesthetic allergy).
* Patients having cesarean section or combined spinal epidural.
* Patients whose epidurals are performed by residents in first month of obstetric rotation and/or having performed fewer than 20 labor epidurals in total.
* Patient needing a translator for procedure.
* Patients who are prisoners.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Time to placement of neuraxial block in parturients with BMI=35-59.9 | Time from start of epidural procedure to placement of epidural needle, not to exceed more than1 hour
  Time period from initially touching the patient's skin to removal of Tuohy needle after catheter placement.
Number of passes to placement of neuraxial block in parturients with BMI=35-59.9 | Time from start of epidural procedure to placement of epidural needle, not to exceed more than1 hour
  Number of times the epidural needle is removed from skin and re-entered

CONTACTS AND LOCATIONS:
Overall Officials: Regina Fragneto, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No